CLINICAL TRIAL: NCT05721612
Title: Evaluation of the Use of Titanium Platelet-rich Fibrin in Sinus Floor Elevation Through Flapless Transcrestal Approach ( a Randomized Controlled Clinical Trial)
Brief Title: Titanium Platelet-rich Fibrin in Sinus Floor Elevation Through Flapless Transcrestal Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPRF_2021
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Sinus Floor Elevation
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental)
  Interventions: Other: Flapless transcrestal sinus lift approach with TPRF
- Control gorup (Active Comparator)
  Interventions: Other: Flapless transcrestal sinus lift approach with PRF

INTERVENTIONS:
Other: Flapless transcrestal sinus lift approach with TPRF — Including 8 patients who will be treated by flapless transcrestal sinus floor elevation using the TPRF as a sole grafting material.
  Arms: Study group
Other: Flapless transcrestal sinus lift approach with PRF — Including 8 patients who will be treated by flapless transcrestal sinus floor elevation using the PRF as a sole grafting material.
  Arms: Control gorup

SUMMARY:
Dental implant therapy in the posterior maxilla may be difficult owing to limited bone height after dental extraction with sinus pneumatization. Several approaches for sinus floor elevation have been documented, and hence flapless transcrestal sinus floor elevation is minimally invasive technique which is used in moderately defected maxilla.

Aim of the study: to evaluate both clinical and radiographic outcomes in sinus floor elevation following dental implant placement using flapless transcrestal sinus lift approach with Titanium platelet rich fibrin (TPRF) as a sole sinus graft material compared to Platelet rich fibrin (PRF).

ELIGIBILITY:
Inclusion Criteria:

* Patient seeking replacement of a missed maxillary posterior teeth by a delayed dental implant procedure.
* Residual bone height is (4-7) mm measured from crestal bone to sinus floor.
* Good oral hygiene

Exclusion Criteria:

* Uncontrolled Diabetes.
* Coagulation disorders.
* Immunological disorders.
* Previous radiation of the head and neck region.
* Abnormal bone physiology.
* Therapy with Bisphosphonates.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Change in bone density | Baseline and 6 months
  Cuts of CBCT (cross sectional, axial and sagittal view), bone density, will be analyzed using On-demand software. The radiographic evaluation will be based on radiological parameters, using reference points and lines at T0 and T1.

SECONDARY OUTCOMES:
Change in implant stability | Baseline and 6 months
  Secondary implant stability will be measured 6 months post-operatively using Osstell device.
change in pain scores | 1st day, 3rd day and 1 week
  Pain (by Visual Analogous Scale) ranges from 0 to 10 0 - No pain. 2 to 4 - Mild pain. 5 to 7 - Moderate pain. 8 to 10 - severe pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt